CLINICAL TRIAL: NCT04865367
Title: To Investigate How Secreted-embryo-derived Trypsin Initiates, Maintains and Terminates Ca2+ (Intracellular Calcium) Signals in Uterine Epithelial Cells
Brief Title: How Secreted-embryo-derived Trypsin Initiates, Maintains and Terminates Ca2+ Signals in Uterine Epithelial Cells
Acronym: Ca2+
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Collaborators: University Women's Hospital Tübingen (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Other Study IDs: 2012-ABU-014-BL
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Infertility; Infertility, Female; Aneuploidy
Keywords: IVF; RNA; Ca2+; embryo; media
MeSH Terms: conditions — Infertility; Infertility, Female; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DEG n1: euploid medium: culture media derived from euploid embryos
  Interventions: Other: Exposure to culture media
- DEG n2: aneuploid medium: culture media derived from aneuploid embryos
  Interventions: Other: Exposure to culture media
- DEG n3: medium arrested embryos: culture media derived from arrested embryos
  Interventions: Other: Exposure to culture media
- DEG n4: control culture medium: pure culture media without contact to embryos
  Interventions: Other: Exposure to culture media

INTERVENTIONS:
Other: Exposure to culture media — Exposure to culture media

SUMMARY:
To develop a deeper understanding of endometrial-embryo crosstalk through basic research, uncover therapeutic targets and to improve reproductive outcome.

DETAILED DESCRIPTION:
Pregnancy is a complex and highly coordinated physiological process that involves implantation of a hatched blastocyst into a decidualizing endometrium. The main purpose of implantation is to ensure that the blastocyst firmly anchors into the decidual stroma, which allows further development by enabling placentation. Although a multitude of cellular events and molecular pathways involved in embryo-uterine crosstalk have been identified in mouse models, a comprehensive understanding of human embryo-uterine interaction is still missing. Our work indicates that endometrial epithelial Ca2+ signalling in response to serine proteases released by human embryos plays an important role in maternal recognition and selection of the conceptus at implantation. Previous studies have demonstrated that trophoblast spheroids can elevate [Ca2+]i in human uterine epithelial cell line (Ishikawa) by activating Ca2+ entry via mechano-sensitive Ca2+ permeable channels leading to the induction of epithelial adhesiveness. However, the mechanism(s) mediating the protease-induced [Ca2+]i transients in human uterine epithelium have not been studied to date. Investigators hypothesise that Na+ entry into the intravillous space via trypsin-activated ENaC will depolarise the cellular membrane and increase [Na+]v sufficiently high to reverse the sodium/calcium exchanger providing means for Ca2+ entry into the intravillous space. Ca2+ diffusion from the microvilli into the bulk cytoplasm will increase [Ca2+]i and, in parallel with SOCE, act as a source for re-filling of the ER. Increased [Ca2+]i will also activate the BK channels leading to repolarisation and termination of Ca2+ entry via the NCX.

By using spent medium from embryos, which will undergo pre-implantation genetic testing, it will become possible to determine, whether the above mentioned mechanisms are influenced by the ploidy status of the embryo.

ELIGIBILITY:
Inclusion Criteria:

* Couples with primary / secondary infertility who are planned to undergo ICSI treatment with PGT-A
* Age of each partner above 18 years

Exclusion Criteria:

* Couples with consanguinity (couple who is 1st or 2nd degree cousins)
* Couples in whom the female partner has a history of:
* Chemotherapy or radiation which impacts the ovarian reserve
* Surgery at the ovaries / adnex region
* Endometriosis
* Couples in whom the male partner has a history of:
* Chemotherapy / Radiation which impacts the semen result
* Surgery at the testicles
* Vasectomy
* Surgery for reversal of vasectomy
* Semen obtained by fine needle aspiration (FNA) or Testicular sperm extraction (TESE)

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female arab
Study Population: Arab ethnicity, with primary / secondary infertility, who undergo an ICSI treatment with preimplantation genetic testing for aneuploidies.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change in markers of protein | 1 day
  Change in markers of protein (PAR2, (p) and SGK1, NFkB, ORAI1-3 and STIM1-2 and COX2) using Western blotting
Change in peak and slope levels of intracellular calcium | 1 day
  Change in peak and slope levels of intracellular calcium
Change in morphohology of cells after incubation with embryo media | 1 day
  Change in morphohology of cells after incubation with embryo media

SECONDARY OUTCOMES:
Performance of ICSI | 1 day
  Defined on day 0 as the number of injected oocytes/number of COCs assigned to the ICSI group
Embryo quality on day 3 | 1 day
  Defined by the number of blastomeres and their division pattern, fragmentation, presence of compaction, vacuoles, granulation and nuclei
Embryo quality on day 5 (Gardner and Schoolcraft,1999) | 1 day
  Gardner and Schoolcraft,1999) defined by:
  * The expansion stage of the blastocyst
  * Quality of the ICM and TE
  * Day on which the biopsy is performed (day 5,6 or 7)
  * Pregnancy outcomes (miscarriages/ectopic pregnancy/neonatal outcome)

CONTACTS AND LOCATIONS:
Overall Officials: BARBARA LAWRENZ, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Dey SK. Roadmap to embryo implantation: clues from mouse models. Nat Rev Genet. 2006 Mar;7(3):185-99. doi: 10.1038/nrg1808. PMID 16485018
- [Background] Kaneko Y, Day ML, Murphy CR. Integrin beta3 in rat blastocysts and epithelial cells is essential for implantation in vitro: studies with Ishikawa cells and small interfering RNA transfection. Hum Reprod. 2011 Jul;26(7):1665-74. doi: 10.1093/humrep/der128. Epub 2011 Apr 30. PMID 21531996
- [Background] Mertzanidou A, Wilton L, Cheng J, Spits C, Vanneste E, Moreau Y, Vermeesch JR, Sermon K. Microarray analysis reveals abnormal chromosomal complements in over 70% of 14 normally developing human embryos. Hum Reprod. 2013 Jan;28(1):256-64. doi: 10.1093/humrep/des362. Epub 2012 Oct 9. PMID 23054067
- [Background] Teklenburg G, Salker M, Heijnen C, Macklon NS, Brosens JJ. The molecular basis of recurrent pregnancy loss: impaired natural embryo selection. Mol Hum Reprod. 2010 Dec;16(12):886-95. doi: 10.1093/molehr/gaq079. Epub 2010 Sep 16. PMID 20847090
- [Background] Quenby S, Vince G, Farquharson R, Aplin J. Recurrent miscarriage: a defect in nature's quality control? Hum Reprod. 2002 Aug;17(8):1959-63. doi: 10.1093/humrep/17.8.1959. PMID 12151421
- [Background] Aplin JD. Embryo implantation: the molecular mechanism remains elusive. Reprod Biomed Online. 2006 Dec;13(6):833-9. doi: 10.1016/s1472-6483(10)61032-2. PMID 17169205
- [Background] Zhang S, Lin H, Kong S, Wang S, Wang H, Wang H, Armant DR. Physiological and molecular determinants of embryo implantation. Mol Aspects Med. 2013 Oct;34(5):939-80. doi: 10.1016/j.mam.2012.12.011. Epub 2013 Jan 2. PMID 23290997
- [Background] Ruan YC, Guo JH, Liu X, Zhang R, Tsang LL, Dong JD, Chen H, Yu MK, Jiang X, Zhang XH, Fok KL, Chung YW, Huang H, Zhou WL, Chan HC. Activation of the epithelial Na+ channel triggers prostaglandin E(2) release and production required for embryo implantation. Nat Med. 2012 Jul;18(7):1112-7. doi: 10.1038/nm.2771. PMID 22729284
- [Background] Rossier BC, Stutts MJ. Activation of the epithelial sodium channel (ENaC) by serine proteases. Annu Rev Physiol. 2009;71:361-79. doi: 10.1146/annurev.physiol.010908.163108. PMID 18928407
- [Background] Marunaka Y, Niisato N. Effects of Ca(2+) channel blockers on amiloride-sensitive Na(+) permeable channels and Na(+) transport in fetal rat alveolar type II epithelium. Biochem Pharmacol. 2002 Apr 15;63(8):1547-52. doi: 10.1016/s0006-2952(02)00880-8. PMID 11996897
- [Background] Salker MS, Hosseinzadeh Z, Alowayed N, Zeng N, Umbach AT, Webster Z, Singh Y, Brosens JJ, Lang F. LEFTYA Activates the Epithelial Na+ Channel (ENaC) in Endometrial Cells via Serum and Glucocorticoid Inducible Kinase SGK1. Cell Physiol Biochem. 2016;39(4):1295-306. doi: 10.1159/000447834. Epub 2016 Sep 8. PMID 27606670
- [Background] Singh Y, Shi X, Zhang S, Umbach AT, Chen H, Salker MS, Lang F. Prolyl hydroxylase 3 (PHD3) expression augments the development of regulatory T cells. Mol Immunol. 2016 Aug;76:7-12. doi: 10.1016/j.molimm.2016.06.003. Epub 2016 Jun 19. PMID 27331863
- [Background] Heijnen EM, Eijkemans MJ, De Klerk C, Polinder S, Beckers NG, Klinkert ER, Broekmans FJ, Passchier J, Te Velde ER, Macklon NS, Fauser BC. A mild treatment strategy for in-vitro fertilisation: a randomised non-inferiority trial. Lancet. 2007 Mar 3;369(9563):743-749. doi: 10.1016/S0140-6736(07)60360-2. PMID 17336650
- [Background] Brosens JJ, Salker MS, Teklenburg G, Nautiyal J, Salter S, Lucas ES, Steel JH, Christian M, Chan YW, Boomsma CM, Moore JD, Hartshorne GM, Sucurovic S, Mulac-Jericevic B, Heijnen CJ, Quenby S, Koerkamp MJ, Holstege FC, Shmygol A, Macklon NS. Uterine selection of human embryos at implantation. Sci Rep. 2014 Feb 6;4:3894. doi: 10.1038/srep03894. PMID 24503642
- [Background] Turco MY, Gardner L, Hughes J, Cindrova-Davies T, Gomez MJ, Farrell L, Hollinshead M, Marsh SGE, Brosens JJ, Critchley HO, Simons BD, Hemberger M, Koo BK, Moffett A, Burton GJ. Long-term, hormone-responsive organoid cultures of human endometrium in a chemically defined medium. Nat Cell Biol. 2017 May;19(5):568-577. doi: 10.1038/ncb3516. Epub 2017 Apr 10. PMID 28394884